CLINICAL TRIAL: NCT05706454
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multi- Centre, Adaptive Phase 2/Phase 3 Study To Evaluate The Efficacy And Safety Of Ramatroban Along With The Standard Of Care In Subjects Hospitalized For SARS-CoV-2 Infection
Brief Title: Phase 2/Phase 3 Study To Evaluate The Efficacy And Safety Of Ramatroban Along With The Standard Of Care In Subjects Hospitalized For COVID Pneumonia
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: KARE Biosciences (Industry)
Collaborators: JSS Medical Research Inc. (Industry); Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Open Philanthropy (Other); Charak Laboratories India Pvt. Ltd (Unknown); Charak Foundation (Unknown); BioLink Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAMBAN-1
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 Pneumonia; COVID-19 Respiratory Infection
Keywords: COVID-19; Ramatroban; Post-Acute Sequelae SARS-CoV-2 infection (PASC); Thromboxane; Prostaglandin D2; F2-Isoprostane
MeSH Terms: conditions — COVID-19 | interventions — ramatroban

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Group, Placebo Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, Investigator and Outcome Assessor Blinded Method of concealment: Pharmacy-controlled Randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ramatroban 75 mg tablet (Experimental)
  Interventions: Drug: Ramatroban
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramatroban — Route of Administration: Oral Dose: 75 mg; Frequency: Twice daily; Total duration of intervention: 28 days.
  Subjects will be evaluated over a study period of approximately 365 days.
  Other Names: BAYu3405; IUPAC Name: 3-[(3R)-3-[(4-fluorophenyl)sulfonylamino]-1,2,3,4-tetrahydrocarbazol-9-yl]propanoic acid
  Arms: Ramatroban 75 mg tablet
Drug: Placebo — Matching placebo will be administered orally twice a day
  Arms: Placebo

SUMMARY:
Phase II/Phase III study to evaluate the safety and efficacy of Ramatroban 75 mg tablet against Placebo in subjects hospitalized for pneumonia due to SARS-CoV-2 infection.

Approximately 324 eligible subjects will be randomized in a 1:1 ratio to one of the two treatment groups.

Group I: Ramatroban 75 mg tablet + Standard of care; Group II: Placebo + Standard of care.

Phase 2

Primary Objective:

To evaluate the safety of Ramatroban 75 mg tablet with the standard of care against Placebo with the standard of care in COVID-19 hospitalized subjects.

Secondary Objective:

To assess the efficacy of Ramatroban 75 mg tablet with the standard of care against Placebo with the standard of care in COVID-19 hospitalized subjects.

Phase 3

Primary Objective:

To evaluate the efficacy of Ramatroban 75 mg tablet with the standard of care against Placebo with the standard of care in COVID-19 hospitalized subjects.

Secondary Objective:

To evaluate the safety of Ramatroban 75 mg tablet with the standard of care against Placebo with the standard of care in COVID-19 hospitalized subjects.

Long COVID [Follow-up Phase- Objectives- (Phase 2 & 3)]

1. To examine lipid mediators, specifically thromboxane A2, prostaglandin D2, F2-isoprostane and/or their metabolites in convalescent subjects after treatment.
2. To assess the efficacy of Ramatroban administered during the acute illness in preventing/mitigating subsequent development of long COVID / PASC

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects of age 18 years and above.
2. Subject (or legally authorized representative) willing to provide informed consent and agrees to comply with planned study procedures.
3. Subjects hospitalized for SARS-COV-2 infection, having hypoxemia (SpO2: ≤ 93% on room air) and radiological evidence supporting COVID-19 pneumonia.
4. Subjects meeting 8-point WHO Ordinal Scale 5 or 6
5. Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR or other commercial or public health assay in any specimen, as documented by either of the following:

   1. PCR positive in a sample collected < 72 hours prior to randomization; OR
   2. PCR positive in sample collected ≥ 72 hours but < 10 days prior to randomization AND non-improving or progressive disease suggestive of ongoing SARS-CoV-2 infection.

   i. Note: In case if the subject is not having previous reports, a quantitative analysis will be performed
6. Women of childbearing potential must agree to either abstinence or use at least one primary form of contraception not including hormonal contraception from the time of screening through Day 36.
7. Agrees to not participate in another clinical trial (both pharmacologic and other types of interventions) for the treatment of COVID-19 through-out the study period

Exclusion Criteria:

1. Subject with immediately life-threatening SARS-CoV-2 infection.

   -Life-threatening disease is defined as respiratory failure, septic shock, and/or multiple organ dysfunction or failure
2. Subjects on invasive mechanical ventilation at screening or randomization.
3. Female subject who is pregnant, breastfeeding, or planning to become pregnant.
4. Subject having other clinically significant gastrointestinal (GI) disease/ GI surgery that in the opinion of the investigator would interfere with the absorption of Ramatroban or subject is unable to swallow oral medications.
5. Subject with pre-existing clinically significant spontaneous bleeding abnormality, or any other condition as per investigator's judgment.
6. Known HIV/Hepatitis B or Hepatitis C infection.
7. Severe liver disease (ALT, AST >5 times the upper limit of normal, total bilirubin > 2 times the upper limit of normal).
8. Subject with known severe renal impairment (estimated glomerular filtration rate ≤30 mL/min/1.73 m2) or receiving continuous renal replacement therapy, hemodialysis, peritoneal dialysis.
9. Subject participated in any other clinical study using any investigational drug in the past 30 days before the screening visit.
10. Subject with a history of life-threatening neoplasms within 5 years prior to the screening visit, other than carcinoma in situ of the cervix or basal cell carcinoma of the skin.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Serious Adverse Events (SAE) | Baseline - Day 29
Time to Clinical recovery (TTCR) | Baseline - Day 15

SECONDARY OUTCOMES:
Composite endpoint of death or need for mechanical ventilation or ECMO | Baseline - Day 29
Rate of mechanical ventilation or vasopressor therapy, or ECMO | Day 29
Ventilator free days | Baseline-Day 29
Duration of hospitalization | Baseline-Day 29
Duration of ICU stay | Baseline-Day 29
Number of subjects who had thrombotic events | Within Day 29
Mortality rate | Till Day 29
Change in hemoglobin, platelets, WBC, creatinine, need for renal replacement. | Baseline- Day 29
Occurrence of serious ventricular arrhythmia | censored at hospital discharge
Total red blood cell units transfused | Baseline -Day 29
Major or Clinically Significant Non-Major Bleeding | Baseline -Day 29
Change from baseline of inflammation and coagulation markers | Baseline- Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gupta, MD, Principal Investigator — KARE Biosciences; Martin Ogletree, PhD, Study Director — Points & Assists, LLC.; Deanna J Nelson, PhD, Study Director — BioLink Life Sciences, Inc.
Locations (7):
- India (7):
  - DEC Health Care, Nellore, Andhra Pradesh
  - Shakti Superspecialty Hospital, Ahmedabad, Gujarat
  - Lifecare Hospital, Mumbai, Maharashtra
  - Sangvi Multispecialty Hospital Pvt Ltd, Pune, Maharashtra
  - Saikrupa Hospital, Pune, Maharashtra
  - Spandan Hospital, Pune, Maharashtra
  - PDEA'S Ayurved Rugnalaya & Sterling Multispeciality Hospital, Pune, Maharashtra